CLINICAL TRIAL: NCT06303349
Title: Predictive Model for the Occurrence of Cerebral Vasospasm Complicating Subarachnoid Haemorrhage by Combined Analysis of the Kinetics of a Panel of Biomarkers.
Acronym: CVSBIODIAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2023/45
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Vasospasm
Keywords: subarachnoid hemorrhage; Cerebral Vasospasm; biomarker; S100 β; IL-6; NSE
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage

STUDY DESIGN:
Intervention Model Description: Prospective single-centre cohort study with prognostic aim, carried out in the neuro-resuscitation unit of the Bordeaux University Hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental arm (Experimental): Patients with subarachnoid hemorrhage, whether aneurysmal or non-aneurysmal, who were admitted to the neuro-resuscitation unit within four days of onset.
  Diagnosis was based on clinical presentation and confirmed by brain imaging
  Interventions: Other: Samples collection

INTERVENTIONS:
Other: Samples collection — from D1 to D10, 1 SSTII (Serum separator tubes II) dry tube of 6 mL blood and 1 EDTA (Ethylenediamine tetraacetic acid) tube of 6 mL blood are collected.
  1 SSTII dry tube of 6 mL cerebral spinal fluid will be collected distally in external ventricular drain, after eliminating the dead volume of the collection burette, for patients with it.

SUMMARY:
The objective is to create a dynamic clinical prediction model that includes routinely measured care and biological biomarkers to predict cerebral vasospasm within 14 days of bleeding in patients treated in the neurosurgical intensive care unit for subarachnoid hemorrhage.

Patients admitted to intensive care will be followed for up to 14 days (D14 time horizon of interest), or until discharge from intensive care if earlier.

Blood samples will be taken from D1 to D10 to isolate the blood biomarkers of interest for each patient.

The measurement of biomarkers and cerebral vasospasm will be blinded to each other.

DETAILED DESCRIPTION:
Subarachnoid hemorrhage (SAH) is the rupture of a cerebral aneurysm, resulting in bleeding into the subarachnoid space.

This condition has significant morbidity and mortality. The patient's functional outcome is primarily determined by the severity of cerebral ischemic lesions that develop during the first few weeks after the acute phase. The main focus of resuscitation management in patients are the 'delayed ischemic lesions'. These lesions are caused by various phenomena, with vasospasm being the most common mechanism. The caliber of cerebral arteries will shrink, reducing the blood flow delivered to the parenchyma, leading to a deficit of energy metabolites in neurons and causing their death. This complication typically occurs within a well-defined time frame, ranging from 3 to 21 days after bleeding, and peaking around the seventh day.

The objective of this study is to create a novel predictive method for symptomatic vasospasm. This method will incorporate routine clinical and radiological biomarkers, as well as innovative biological assays. The aim is to enable earlier diagnosis and even pre-emptive treatment of this pathology.

Several studies have examined the predictive potential of various blood biomarkers for neurological prognosis and the incidence of delayed brain damage in patients. These studies have demonstrated strong associations between them. For instance, one study found that patients with the most severe vasospasm had a significantly higher peak in cerebrospinal fluid of several biomarkers associated with neurodegeneration, such as Neuron Specific Enolase (NSE). Additionally, the plasma concentration-time curves demonstrated simultaneous elevations during periods of vasospasm.

However, no study has examined the practical clinical use of these biomarkers during hospitalization to predict the occurrence of vasospasm on a daily basis or at specific times of interest. This is particularly important as the pathophysiological time sequence appears to be common to all patients. A single study has attempted to establish a predictive algorithm for delayed cerebral lesions, achieving a certain degree of effectiveness (over 90% correct predictions and sensitivity of around 93%), by combining a single biomarker assay and clinical parameters. However, this study only focuses on ischemic lesions at 6 weeks and cannot be used to guide therapy during initial management.

Within the framework of a predictive statistical model, the investigators wish to study the possibility of combining routine clinical and radiological parameters with iterative assays of a panel of biomarkers covering several pathophysiological pathways (which would be easily assayable in the plasma of all patients) to predict on a daily basis (or at certain times of clinical interest) the risk of occurrence of cerebral vasospasm, with a view to being able to trigger diagnostic (or even therapeutic) procedures during initial management to prevent the ischemic cascade.

To this end, the investigators have chosen 3 assays as a priority, targeting three previously described pathophysiological pathways.

For neuroinflammation :

* Interleukin-6 (IL-6)

For cerebral cellular damage:

* Neuron Specific Enolase (NSE)
* The β-subunit of the S100 protein (S100 β)

To enable this prediction, the investigators propose to use an innovative statistical method in the health sciences. Repeated biomarker assays can be integrated into complex event prediction models: the joint modeling of a longitudinal data model, for estimating individual biomarker trajectories over time, and a survival model, for estimating event risk with the current value or slope of the biomarker, enables precise event prediction. These models enable either static prediction (at a given time horizon) or dynamic prediction (with re-estimation of risk during follow-up). They also allow the concomitant integration of several biomarkers. Lastly, a model estimated on the study population could be transposed to other populations, thus making it possible to obtain risk models for this event.

The aim of this research is to develop tools for daily clinical prediction of the onset of symptomatic vasospasm, using routine clinical and radiological parameters as well as innovative biological assays, with a view to triggering earlier diagnostic and even therapeutic responses than with the usual screening methods, which are severely limited and not always usable.

ELIGIBILITY:
Inclusion Criteria:

* Subarachnoid hemorrhage (of aneurysmal or non-aneurysmal etiology) less than 4 days prior to admission to neuro-resuscitation, diagnosed on clinical presentation and confirmed by brain imaging.
* Free, informed and written consent signed by the patient (or, failing this, his or her representative).
* Patient entitled to or affiliated with social security

Exclusion Criteria:

* Significant vasospasm on admission to the department, diagnosed on initial imaging
* Patient whose short-term survival (48 hours) appears compromised
* Contraindication to perfusion CT scan
* Pregnant or breast-feeding women
* Patient under legal protection (persons deprived of liberty or under guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Occurrence of cerebral vasospasm | Day 14 after inclusion
  Occurrence of cerebral vasospasm within 14 days of ICU (Intensive Care Unit) admission.

SECONDARY OUTCOMES:
Biomarkers measurements | Day 10 after inclusion
  Daily Serum measurements of the following markers from D1 to D10:
  * IL-6
  * NSE
  * S100 β
WFNS (World Federation of Neurologic Surgeons) score | up to Day 10 after inclusion
  Initial WFNS score : From grade I (13% of bad evolution at 6 months) to grade V (68% of bad evolution à 6 months)
Glasgow score | up to Day 10 after inclusion
  Hourly Glasgow score (scale from 3 :deep coma to 15 : fully conscious)
Medical Research Council (MRC) score | up to Day 10 after inclusion
  Presence and intensity (MRC score) of motor deficit. scale from 0 : no movement is observed to 5 : full range of motion
PtiO2 (oxygen pressure in the cerebral tissue) | up to Day 10 after inclusion
  Hourly PtiO2 data.
Transcranial Doppler | up to Day 10 after inclusion
  Daily transcranial Doppler data from D1 to D10;
Modified Fisher score | up to Day 10 after inclusion
  Modified Fisher score from initial imaging. Scale from 0(no subarachnoid hemorrhage / no intraventricular hemorrhage / incidence of symptomatic vasospasm: 0%) to 4 (thick subarachnoid hemorrhage / intraventricular hemorrhagepresent /the incidence of symptomatic vasospasm: 40%)
Non-significant angiographic vasospasm | up to Day 10 after inclusion
  Presence of non-significant angiographic vasospasm on initial diagnostic/therapeutic arteriography or on follow-up imaging from D1 to D10.
Non-significant perfusion anomaly | up to Day 10 after inclusion
  Presence of a non-significant perfusion anomaly on follow-up imaging from D1 to D10.
Glasgow Outcome Scale -Extended (GOS-E) | up to Day 14 after inclusion
  GOS-E at ICU discharge. 8 levels (1 to 8) are in the scale: Minimum Score = 1 : Dead Maximum Score = 8 : Upper Good Recovery
Cerebral ischemic lesions | up to Day 14 after inclusion
  Presence of delayed cerebral ischemic lesions on last imaging before discharge.
Occurrence of symptomatic vasospasm | up to Day 14 after inclusion
  Occurrence of symptomatic vasospasm in non-severe SAH during ICU stay.
Organ infection | up to 10 days after inclusion
  The occurrence of an organ infection diagnosed according to the Centers for Disease Control and Prevention/National Healthcare Safety Networkdefinition associated with the initiation of antibiotic therapy.
Severe pneumonia | up to 10 days after inclusion
  The occurrence of severe pneumonia within the first 10 days of the intensive care unit stay
Septic shock | up to 10 days after inclusion
  The occurrence of septic shock within the first 10 days of the intensive care unit stay

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire CANE, Dr, Principal Investigator — University Hospital, Bordeaux; Hugues De COURSON, Dr, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France